CLINICAL TRIAL: NCT03819699
Title: Interventional, Open-label, Multiple-immunisation Study of the Immunogenicity, Pharmacodynamics and Safety of Lu AF20513 in Patients With Mild Alzheimer's Disease or Mild Cognitive Impairment Due to Alzheimer's Disease
Brief Title: Study With Lu AF20513 in Patients With Mild Alzheimer's Disease (AD) or Mild Cognitive Impairment (MCI) Due to AD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: New data: The study was terminated based on new efficacy data from another study
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18086A
Record Dates: First submitted 2019-01-25; First posted 2019-01-28 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 - dose regimen 1 (Experimental): Cohort 1: encompasses patients enrolled prior to the PA1
  Interventions: Drug: Lu AF20513
- Cohort 2 - dose regimen 2 (Experimental): Cohort 2: 10 patients who will receive one administration of booster vaccine prior to the first IMP administration
  Interventions: Drug: Lu AF20513; Biological: booster vaccine
- Cohort 2 - dose regimen 3 (Experimental): Cohort 2: 10 patients who will not receive a booster vaccine
  Interventions: Drug: Lu AF20513

INTERVENTIONS:
Drug: Lu AF20513 — Lu AF20513 suspension for injection
Biological: booster vaccine — booster vaccine (Cohort 2) - to be administered as per national recommendations
  Arms: Cohort 2 - dose regimen 2

SUMMARY:
The purpose of this study is to study the effect of monthly dosing with a single dose of Lu AF20513, with and without booster vaccine, on antibody response.

DETAILED DESCRIPTION:
Cohort 1 encompasses 8 patients enrolled prior to the Protocol Amendment (PA) 1, dose regimen 1.

Cohort 2 includes patients enrolled under the PA and will consist of 20 patients, randomly assigned to two arms:

* dose regimen 2: 10 patients who will receive one administration of booster vaccine 4 weeks prior to the first IMP administration
* dose regimen 3: 10 patients who will not receive a booster vaccine

After the PA1, the study consists of the following periods:

* Screening Period - up to 12 weeks
* Priming period: 28 weeks, monthly dosing with Lu AF20513
* Maintenance Period - 56 weeks, quarterly dosing with Lu AF20513
* Follow-up Period - 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* The patient has a diagnosis of AD or Mild Cognitive Impairment (MCI) due to AD.
* The patient has evidence of an abnormal amyloid and tau status, consistent with AD, by means of a positive CSF test at screening
* The patient is aged ≥50 and ≤85 years. If a woman, the patient must be post-menopausal.

Exclusion Criteria:

* The patient has participated in a clinical study where he/she has received passive or active anti-Aβ immunotherapy or other active immunisation for the treatment of AD.
* The patient has, in the investigator's opinion, evidence and/or history (clinically or on MRI) of any clinically significant neurodegenerative disease, serious neurological disorder, other intracranial or systemic diseases or conditions resulting in a definite or probable diagnosis of Major or Mild Neuro-Cognitive disorder other than AD, per DSM-5® criteria.

Other in- and exclusion criteria may apply

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
AUC | From Week 0 to Week 28
  Area under antibody titre curve (AUC) induced upon treatment with Lu AF20513
Cmax | From Week 0 to Week 28
  maximum antibody titre (Cmax) induced upon treatment with Lu AF20513
Titre response | From Week 0 to Week 28
  Any patients with antibody titre above the patient's baseline titre in either of the applied assays for antibody assessment

SECONDARY OUTCOMES:
Amyloid load | From baseline to week 84
  Change in composite cortical standard uptake volume ratio based on PET scans (amyloid PET-SUVR)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (3):
- Finland (2):
  - University of Eastern Finland, Brain Research Unit (FI002), Kuopio
  - Clinical Research Services Turku Oy (FI001), Turku
- Karolinska University Hospital, Huddinge (SE001), Stockholm, Sweden